CLINICAL TRIAL: NCT05944640
Title: Dynamic Parameters of Glucose Control in Relation to Biomarkers in Serum and Intraocular Fluid in Diabetic Patients With Ocular Complications
Brief Title: Dynamic Parameters of Glucose Control in Relation to Biomarkers in Serum and Intraocular Fluid in Patients With Diabetes
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Czech Health Research Council (Unknown)
Responsible Party: Principal Investigator, Martin Prázný, Prof., Charles University, Czech Republic
Other Study IDs: NU22-01-00077
Record Dates: First submitted 2023-02-07; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Complications
Keywords: biomarkers; retinopathy; miRNA; diabetes mellitus; glucose variability
MeSH Terms: conditions — Diabetes Complications; Retinal Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We determined the biomarkers that are present in blood and/or intraocular fluid of patients with ocular complications. MicroRNA (miRNA) and inflammatory chemokines/cytokines (VEGF, IL-6, IL-8, TNF-α, IL-1β and MCP-1) are the candidates. miRNA are small non-coding RNAs, which regulate gene expression at the post-transcriptional level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with DR: Adult patients with T1DM or T2DM with any form of diabetic retinopathy and diabetic macular edema, indicated for ocular surgical procedure as standard of care. Blood samples and samples of intraocular fluids will bee taken during the ocular surgery.
  Interventions: Procedure: Intraocular surgery
- Patients without DR: Adult patients with T1DM or T2DM without any signs of diabetic retinopathy, indicated for ocular surgical procedure from other reasons as standard of care. Blood samples and samples of intraocular fluids will bee taken during the ocular surgery.
  Interventions: Procedure: Intraocular surgery
- Control group: Subjects without diabetes mellitus indicated for ocular surgery from other reasons (cataract, retinal detachment, macular hole, idiopathic epiretinal membrane) as standard of care. Blood samples and samples of intraocular fluids will bee taken during the ocular surgery.
  Interventions: Procedure: Intraocular surgery

INTERVENTIONS:
Procedure: Intraocular surgery — Pars plana vitrectomy or cataract surgery.

SUMMARY:
Our project investigates the new characteristics of diabetic retinopathy using liquid eye biopsy in combination with novel parameters of glucose control obtained with continuous glucose monitoring. This approach will bring new knowledge and implications for future therapies.

DETAILED DESCRIPTION:
Diabetic retinopathy is one of the most common causes of blindness in developed countries. The short-term glucose fluctuations have been suggested as a factor contributing to the risk of diabetic complications including ocular complications. We hypothesize that modulatory and other biological abilities of miRNAs and inflammatory chemokines/cytokines have a significant impact on the development and the progression of diabetic retinopathy. Our main goal is to identify the biomarkers that will in time be used for new screening, diagnostic, and treatment strategies for patients with diabetic retinopathy, bring a better prevention and early treatment to them and thus improve their quality of life while saving the cost associated with advanced forms of retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or type 2 diabetes
* ≥ 18 years old
* treatment with insulin for at least 5 years prior baseline
* any form of diabetic retinopathy and macular edema
* HbA1c < 10%
* written informed consent prior to starting study related activity

Exclusion Criteria:

* any active intraocular or periocular infectious or non-infectious inflammation in study eye
* uncontrolled glaucoma
* history of intraocular inflammation or trauma in study eye
* intravitreal anti-VEGF therapy in study eye during a 3-month perido prior to baseline
* use of corticosteroid intravitreal implant in study eye at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with T1DM or T2DM treated with insulin with or without any form of diabetic retinopathy and the matched controls, who are indicated to ocular surgery procedure as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
miRNA | Year 2025
  miRNA expression measuer by real-time PCR method in plasma and vitreous samples (units: threshold cycle)
TIR | Year 2025
  Percentage of time in target ranges

SECONDARY OUTCOMES:
miRNA expression differences | Year 2025
  miRNA expression differences analysis between diabetic patients with and without diabetic retinopathy (units: fold change)
Glycemic variability | Year 2025
  Expressed as the standard deviation
Mean sensor glucose concentration | Year 2025
  Measured by rtCGM

CONTACTS AND LOCATIONS:
Overall Officials: Martin Prázný, Prof., Principal Investigator — Charles University and General University Hospital in Prague
Locations (1):
- General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ceriello A, Esposito K, Piconi L, Ihnat MA, Thorpe JE, Testa R, Boemi M, Giugliano D. Oscillating glucose is more deleterious to endothelial function and oxidative stress than mean glucose in normal and type 2 diabetic patients. Diabetes. 2008 May;57(5):1349-54. doi: 10.2337/db08-0063. Epub 2008 Feb 25. PMID 18299315
- [Background] Soupal J, Skrha J Jr, Fajmon M, Horova E, Mraz M, Skrha J, Prazny M. Glycemic variability is higher in type 1 diabetes patients with microvascular complications irrespective of glycemic control. Diabetes Technol Ther. 2014 Apr;16(4):198-203. doi: 10.1089/dia.2013.0205. Epub 2014 Jan 8. PMID 24401008
- [Background] Zoppini G, Verlato G, Targher G, Casati S, Gusson E, Biasi V, Perrone F, Bonora E, Muggeo M. Is fasting glucose variability a risk factor for retinopathy in people with type 2 diabetes? Nutr Metab Cardiovasc Dis. 2009 Jun;19(5):334-9. doi: 10.1016/j.numecd.2008.02.007. Epub 2008 Jun 20. PMID 18571393
- [Background] Takao T, Ide T, Yanagisawa H, Kikuchi M, Kawazu S, Matsuyama Y. The effects of fasting plasma glucose variability and time-dependent glycemic control on the long-term risk of retinopathy in type 2 diabetic patients. Diabetes Res Clin Pract. 2011 Feb;91(2):e40-2. doi: 10.1016/j.diabres.2010.10.009. Epub 2010 Oct 29. PMID 21035886
- [Background] Vujosevic S, Aldington SJ, Silva P, Hernandez C, Scanlon P, Peto T, Simo R. Screening for diabetic retinopathy: new perspectives and challenges. Lancet Diabetes Endocrinol. 2020 Apr;8(4):337-347. doi: 10.1016/S2213-8587(19)30411-5. Epub 2020 Feb 27. PMID 32113513
- [Background] Meister G, Landthaler M, Dorsett Y, Tuschl T. Sequence-specific inhibition of microRNA- and siRNA-induced RNA silencing. RNA. 2004 Mar;10(3):544-50. doi: 10.1261/rna.5235104. PMID 14970398
- [Background] Martinez B, Peplow PV. MicroRNAs as biomarkers of diabetic retinopathy and disease progression. Neural Regen Res. 2019 Nov;14(11):1858-1869. doi: 10.4103/1673-5374.259602. PMID 31290435
- [Background] Boss JD, Singh PK, Pandya HK, Tosi J, Kim C, Tewari A, Juzych MS, Abrams GW, Kumar A. Assessment of Neurotrophins and Inflammatory Mediators in Vitreous of Patients With Diabetic Retinopathy. Invest Ophthalmol Vis Sci. 2017 Oct 1;58(12):5594-5603. doi: 10.1167/iovs.17-21973. PMID 29084332
- [Background] Wu H, Hwang DK, Song X, Tao Y. Association between Aqueous Cytokines and Diabetic Retinopathy Stage. J Ophthalmol. 2017;2017:9402198. doi: 10.1155/2017/9402198. Epub 2017 Jun 7. PMID 28680705
- [Background] Mastropasqua R, D'Aloisio R, Di Nicola M, Di Martino G, Lamolinara A, Di Antonio L, Tognetto D, Toto L. Relationship between aqueous humor cytokine level changes and retinal vascular changes after intravitreal aflibercept for diabetic macular edema. Sci Rep. 2018 Nov 8;8(1):16548. doi: 10.1038/s41598-018-35036-9. PMID 30410092